CLINICAL TRIAL: NCT06869200
Title: A Prospective, Multicenter, Single-Blind, Randomized Controlled Clinical Trial of an Autologous Platelet-Rich Concentrated Growth Factor (CGF) Preparation Kit for the Treatment of Knee Osteoarthritis
Brief Title: Study on the Use of a Concentrated Growth Factor Preparation Kit for the Treatment of Knee Osteoarthritis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Hongzhi Biotechnology Co. (Industry)
Collaborators: Nanfang Hospital, Southern Medical University (Other); Shantou Central Hospital (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HZJKCGFOA202501
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; concentrated growth factors (CGF); platelet-rich plasma; Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC); Intra-articular Injection
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Injections, Intra-Articular

STUDY DESIGN:
Who Masked: Participant
Masking Description: As the primary outcome measure of this study relies on subjective evaluation by the participants, a single-blind design is adopted to avoid bias introduced by participants' evaluations. During the informed consent process, investigators should clearly inform participants that they will be randomly assigned to one of the two treatment groups, but they will not be informed of which group they have been allocated to until the end of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CGF Treatment Group (Experimental): Participants in this arm will receive three intra-articular injections of Concentrated Growth Factor (CGF) prepared using the autologous platelet-rich CGF preparation kit. The injections will be administered at weekly intervals over a period of three weeks.
  Interventions: Device: Concentrated Growth Factor (CGF) Intra-articular Injection
- PRP Treatment Group (Active Comparator): Participants in this arm will receive three intra-articular injections of Platelet-Rich Plasma (PRP) prepared using a disposable PRP preparation device. The injections will be administered at weekly intervals over a period of three weeks.
  Interventions: Device: Platelet-Rich Plasma (PRP) Intra-articular Injection

INTERVENTIONS:
Device: Concentrated Growth Factor (CGF) Intra-articular Injection — Preparation Method: The CGF is prepared using an autologous platelet-rich preparation kit specifically designed to concentrate growth factors from the patient's own blood. The process involves a specialized centrifugation technique that yields a high concentration of growth factors, including platelet-derived growth factor (PDGF), transforming growth factor-beta (TGF-β), and other bioactive molecules.
  Rationale: This intervention leverages the body's natural healing response by utilizing autologous growth factors to enhance the repair of cartilage and other joint tissues affected by osteoarthritis. The high concentration of bioactive molecules in CGF is believed to provide a more potent therapeutic effect compared to other platelet-rich therapies.
  Arms: CGF Treatment Group
Device: Platelet-Rich Plasma (PRP) Intra-articular Injection — Preparation Method: The PRP is prepared using a disposable PRP preparation device that separates and concentrates platelets from the patient's blood. This process enriches the plasma with platelets and associated growth factors.
  Rationale: PRP has been widely used in clinical practice for its ability to promote tissue healing and reduce inflammation in osteoarthritis. It serves as an active comparator in this study, allowing for a direct comparison of the therapeutic efficacy and safety profile of CGF against a well-established treatment modality.
  Arms: PRP Treatment Group

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness and safety of an autologous platelet-rich concentrated growth factor (CGF) preparation kit for the treatment of knee osteoarthritis in patients diagnosed with this condition. The main question it aims to answer is:

Can the CGF preparation kit effectively improve symptoms and reduce pain in patients with knee osteoarthritis compared to a control intervention? Researchers will compare the CGF treatment group to a control group using platelet-rich plasma (PRP) to see if the CGF intervention results in greater improvements in knee function and pain relief.

Participants will:

Undergo three intra-articular injections of CGF or PRP into the knee joint at weekly intervals.

Complete assessments including the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) and Visual Analog Scale (VAS) for pain at specified intervals.

Be monitored for safety and potential adverse events throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, with no gender restrictions;
* Patients diagnosed with knee osteoarthritis according to the "Chinese Guidelines for the Diagnosis and Treatment of Osteoarthritis (2024 Edition)" by the Chinese Osteoarthritis Diagnosis and Treatment Guidelines Expert Group;
* Radiographic evidence of knee osteoarthritis with Kellgren-Lawrence grading of II to IV;
* Visual Analog Scale (VAS) pain score ≥ 4 (moderate or higher pain) and WOMAC score ≥ 24;
* For participants with eligible bilateral knee osteoarthritis, the more severely affected knee will be treated, while the other knee will not be intervened during the study period. If the severity is equal on both sides, the left knee will be selected for intervention;
* The patient or their legal guardian is able to understand the purpose of the study and provide informed consent.

Exclusion Criteria:

* Patients with a confirmed diagnosis of other inflammatory diseases of the knee joint, such as rheumatoid arthritis, psoriatic arthritis, or gouty arthritis; Patients with a confirmed diagnosis of bleeding disorders (e.g., allergic purpura, hemophilia, idiopathic thrombocytopenic purpura), hematologic malignancies (e.g., leukemia), or those with unconfirmed bleeding disorders but coagulation dysfunction (coagulation parameters PT, APTT, INR > 1.5 times the upper limit of normal);
* Patients who have undergone or are planned to undergo knee osteoarthritis surgery within the past 6 months or during the trial period;
* Patients with local infections at the injection site (e.g., septic arthritis, tuberculous arthritis, or local soft tissue infections) or severe systemic infections (e.g., sepsis);
* Patients with untreated malignant diseases such as malignancies, which may interfere with the safety and efficacy assessments of the study and affect the patient's participation in the study;
* Patients with severe hepatic or renal dysfunction [hepatic function indicators alanine aminotransferase (ALT), aspartate aminotransferase (AST) > 2 times the upper limit of normal; renal function indicators serum creatinine (Cr), blood urea nitrogen (BUN) > 2 times the upper limit of normal];
* Patients with hemoglobin < 10 g/dL or platelet count < 125 × 10^9/L;
* Patients who have used any Chinese or Western medications or therapies for the treatment of knee osteoarthritis within 1 week prior to randomization;
* Patients who have received intra-articular injections or related drug therapies within the past 3 months;
* Women who are planning a pregnancy, breastfeeding, or pregnant during the entire clinical study period;
* Patients who have participated in other interventional drug or medical device clinical trials within 1 month prior to enrollment;
* Other situations where the investigator deems the patient unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | One month after the first injection
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is used to assess pain, stiffness, and physical function in patients with hip and knee osteoarthritis. The score ranges from 0 to 96 (using a 5-point Likert scale) or 0 to 240 (using a visual analog scale [VAS]), with lower scores indicating better outcomes.

SECONDARY OUTCOMES:
The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 2 and 3 month after the first injection
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is used to assess pain, stiffness, and physical function in patients with hip and knee osteoarthritis. The score ranges from 0 to 96 (using a 5-point Likert scale) or 0 to 240 (using a visual analog scale [VAS]), with lower scores indicating better outcomes.
The Visual Analog Scale (VAS) | 1，2，and 3 month after the first injection
  The Visual Analog Scale (VAS) is used to measure the intensity of pain experienced by patients. The VAS score ranges from 0 to 10, with lower scores indicating better outcomes (i.e., less pain).

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Nanfang Hospital,, Guangzhou, Guangdong
  - Shantou Central Hospital, Shantou, Guangdong
  - The Third Affiliated Hospital,Sun Yat-Sen University., Guangdong, Guangzhou

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pereira D, Peleteiro B, Araujo J, Branco J, Santos RA, Ramos E. The effect of osteoarthritis definition on prevalence and incidence estimates: a systematic review. Osteoarthritis Cartilage. 2011 Nov;19(11):1270-85. doi: 10.1016/j.joca.2011.08.009. Epub 2011 Aug 24. PMID 21907813
- [Background] Michael JW, Schluter-Brust KU, Eysel P. The epidemiology, etiology, diagnosis, and treatment of osteoarthritis of the knee. Dtsch Arztebl Int. 2010 Mar;107(9):152-62. doi: 10.3238/arztebl.2010.0152. Epub 2010 Mar 5. PMID 20305774
- [Background] Katz JN, Arant KR, Loeser RF. Diagnosis and Treatment of Hip and Knee Osteoarthritis: A Review. JAMA. 2021 Feb 9;325(6):568-578. doi: 10.1001/jama.2020.22171. PMID 33560326
- [Background] Molnar V, Matisic V, Kodvanj I, Bjelica R, Jelec Z, Hudetz D, Rod E, Cukelj F, Vrdoljak T, Vidovic D, Staresinic M, Sabalic S, Dobricic B, Petrovic T, Anticevic D, Boric I, Kosir R, Zmrzljak UP, Primorac D. Cytokines and Chemokines Involved in Osteoarthritis Pathogenesis. Int J Mol Sci. 2021 Aug 26;22(17):9208. doi: 10.3390/ijms22179208. PMID 34502117